CLINICAL TRIAL: NCT03563248
Title: A Randomized Phase 2 Study of Losartan and Nivolumab in Combination With FOLFIRINOX and SBRT in Localized Pancreatic Cancer
Brief Title: Losartan and Nivolumab in Combination With FOLFIRINOX and SBRT in Localized Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry); Stand Up To Cancer (Other); Lustgarten Foundation (Other)
Responsible Party: Principal Investigator, Jennifer Wo, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-179
Record Dates: First submitted 2018-06-07; First posted 2018-06-20 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox; Losartan; Nivolumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- FOLFIRINOX: SBRT: Surgery (Active Comparator): The FOLFIRINOX regimen will be administered intravenously. Treatment will be every 14 days +3/ -1 at physician discretion
  * SBRT should be administered 2-6 weeks after completing chemotherapy
  * All participants will undergo an attempt at definitive surgical resection following SBRT
  Interventions: Drug: FOLFIRINOX; Radiation: SBRT; Procedure: Surgery
- FOLFIRINOX+Losartan:SBRT+Losartan:Surgery (Experimental): The FOLFIRINOX regimen will be administered intravenously. Treatment will be every 14 days +3/ -1 at physician discretion
  * Losartan will be administered orally as a tablet to be taken by the patient at home every day
  * SBRT should be administered 2-6 weeks after completing chemotherapy
  * All participants will undergo an attempt at definitive surgical resection following SBRT
  Interventions: Drug: FOLFIRINOX; Drug: Losartan; Radiation: SBRT; Procedure: Surgery
- FOLFIRINOX+Losartan:SBRT+Nivolumab+Losartan:Sur (Experimental): The FOLFIRINOX regimen will be administered intravenously. Treatment will be every 14 days +3/ -1 at physician discretion
  * Losartan will be administered orally as a tablet to be taken by the patient at home every day
  * SBRT should be administered 2-6 weeks after completing chemotherapy
  * Participants will receive nivolumab during SBRT
  * All participants will undergo an attempt at definitive surgical resection following SBRT
  Interventions: Drug: FOLFIRINOX; Drug: Losartan; Drug: Nivolumab; Radiation: SBRT; Procedure: Surgery
- FOLFIRINOX x 8 : SBRT + Nivolumab : Surgery (Experimental): * The FOLFIRINOX regimen will be administered intravenously. Treatment will be every 14 days +3/ -1 at physician discretion
  * SBRT should be administered 2-6 weeks after completing chemotherapy
  * Participants will receive nivolumab during SBRT
  * All participants will undergo an attempt at definitive surgical resection following SBRT
  Interventions: Drug: FOLFIRINOX; Drug: Nivolumab; Radiation: SBRT; Procedure: Surgery

INTERVENTIONS:
Drug: FOLFIRINOX — FOLFIRINOX is a combination of 4 chemotherapy agents that may help shrink your tumor before surgery
  * 5-Fluorouracil (5-FU) - 400 mg/m2 on day one, followed by 1200 mg/m2 by continuous infusion for the subsequent 46-48 hours
  * Oxaliplatin - 85 mg/m2 by intravenous infusion over 120 minutes on day 1 of each 14 day cycle
  * Irinotecan - administered at a starting dose of 180 mg/m2 by intravenous infusion over 90 minutes on day 1 of each 14 day cycle
  * Leucovorin - Administered at a starting dose of 400 mg/m2 over 2 hours on day 1 of each 14 day cycle
Drug: Losartan — Losartan is a drug that is used to lower blood pressure
  Arms: FOLFIRINOX+Losartan:SBRT+Losartan:Surgery; FOLFIRINOX+Losartan:SBRT+Nivolumab+Losartan:Sur
Drug: Nivolumab — Nivolumab is an antibody that may cause programmed cell death of cancer cells
  Arms: FOLFIRINOX x 8 : SBRT + Nivolumab : Surgery; FOLFIRINOX+Losartan:SBRT+Nivolumab+Losartan:Sur
Radiation: SBRT — Radiation therapy is believed to increase the likelihood of response of immunotherapy
Procedure: Surgery — definitive surgical resection

SUMMARY:
This research study is studying a combination of interventions as a possible treatment for pancreatic tumor.

The interventions involved in this study are:

* FOLFIRINOX which is made up of 4 different drugs:

  * 5-Fluorouracil (5-FU)
  * Oxaliplatin
  * Irinotecan
  * Leucovorin
* Losartan
* Nivolumab
* Radiation Therapy
* Surgery

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has approved FOLFIRINOX as a treatment option for this disease.

The FDA has not approved losartan or nivolumab for this specific disease but they have been approved for other uses.

FOLFIRINOX is a combination of 4 chemotherapy agents that may help shrink your tumor before surgery. Losartan is a drug that is used to lower blood pressure. Nivolumab is an antibody (a cell that attaches to other cells to fight off infection) that may cause programmed cell death of cancer cells. Radiation therapy is believed to increase the likelihood of response of immunotherapy (the prevention/treatment of a disease through an immune response).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed localized pancreatic adenocarcinoma; borderline/potentially resectable or locally advanced.
* Borderline resectable is defined by the NCCN as tumors with venous involvement of the SMV/portal vein demonstrated tumor abutment with or without impingement and narrowing of the lumen, either tumor thrombus or encasement but with suitable vessel proximal and distal to the area of vessel involvement, allowing for safe resection or reconstruction; gastroduodenal artery encasement up to the hepatic artery with either short segment encasement or direct abutment of the hepatic artery, without extension to the celiac axis; or tumor abutment of the SMA not to exceed greater than 180 degrees of the circumference of the vessel wall. Tumors involving retroperitoneal structures that can be surgically removed (i.e. kidney), will also be included.
* Localized is defined as no extrapancreatic disease, no evidence (on CT) of involvement of the celiac axis or SMA, no evidence (CT or MRI) of occlusion of the SMV or SMPV confluence, no evidence of gross peritoneal or distant metastases on staging laparoscopy or laparotomy.
* Locally advanced unresectable disease is defined by the NCCN as: Tumors of the head that have greater than 180 degrees of SMA encasement or any celiac abutment, unreconstructable SMV or portal occlusion, or aortic invasion or encasement. Tumors of the body with SMA or celiac encasement of greater than 180 degrees, unreconstructable SMV or portal occlusion, or aortic invasion. Tumors of the tail with SMA or celiac encasement of greater than 180 degrees. Irrespective of location, all tumors with evidence of nodal metastasis outside of the resection field are deemed unresectable.
* Age > 18 years
* ECOG performance status 0-1
* Baseline Systolic Blood Pressure (SBP) > 100 mm Hg. This is based on the average of two values - separate seated, resting measurements taken five minutes apart. BP does not need to be checked in both arms unless a reading is below 110 mm Hg, in which case the other arm can be checked as well. If BP is checked in both arms, the higher value is deemed accurate for calculating the average.
* Normal organ and marrow function as defined below:

  * absolute neutrophil count ≥ 1,500/mm3
  * platelets ≥ 100,000/mm3
  * total bilirubin ≤ 1.5 x institutional upper limit of normal if no biliary stenting has been done OR 2.0 x upper limit of normal if patient is s/p biliary stenting OR two down trending values
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional upper limit of normal
  * Potassium (not hemolyzed) < 5 mmol/L
  * creatinine ≤ 1.5 mg/ dL OR
  * creatinine clearance ≥ 30 mL/min (as estimated by Cockcroft Gault Equation)
* (140 - age [yrs]) (body wt [kg]) -Creatinine clearance for males = ------------
* (72) (serum creatinine [mg/dL])
* Creatinine clearance for females = 0.85 x male value
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 5 months after the last dose of investigational drug.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab
* Women must not be breastfeeding
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product. Women who are not of childbearing potential, ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception
* Ability to understand and the willingness to sign a written informed consent document
* If applicable, must be on a stable dose of dexamethasone 2 mg or less for 7 days prior to initiation of treatment

Exclusion Criteria:

* NOTE: Patients enrolled to the randomized portion of the study (arms 1 thru 3) may not be already treated on ACE or ARB therapy for hypertension or renal protection (with diabetes) at the time of enrollment. If patients are receiving ACE or ARB therapy, they may ONLY be considered for the exploratory arm, Arm 4.
* Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator), such as significant cardiac or pulmonary morbidity e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months, ongoing infection as manifested by fever.
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test (serum or urine) at baseline. (Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.)
* Any prior chemotherapy, radiation therapy, immunotherapy, or biologic ('targeted') therapy for treatment of the patient's pancreatic tumor
* Treatment for other invasive carcinomas within the last five years who are at greater than 5% risk of recurrence at time of eligibility screening. Carcinoma in-situ and basal cell carcinoma/ squamous cell carcinoma of the skin are allowed.
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* Known, existing uncontrolled coagulopathy
* Prior systemic fluoropyrimidine therapy within the past 10 years. Prior topical fluoropyrimidine use is allowed. Prior unanticipated severe reaction to fluoropyrimidine therapy, or known hypersensitivity to 5-fluorouracil or known DPD deficiency.
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance or oral drug intake.
* Major surgery, excluding laparoscopy, within 4 weeks of the start of study treatment, without complete recovery
* Concomitant use of cimetidine, as it can decrease the clearance of 5-FU. Another H2-blocker or proton pump inhibitor may be substituted before study entry
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 5-fluorouracil, irinotecan, oxaliplatin, or losartan
* Other serious medical conditions that the investigator feels might compromise study participation
* An active, known or suspected autoimmune disease other than those listed below. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* A condition requiring systemic treatment with either corticosteroids (> 15 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 15 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* Known history of active TB (Bacillus Tuberculosis)
* Known positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 5 months for woman and 7 months for men, after the last dose of trial treatment.
* Known history of, or any evidence of active, non-infectious pneumonitis
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* History of severe hypersensitivity reaction to any monoclonal antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with R0 resection | Up to 8 months after baseline
  R0 resection is defined as microscopically negative margins determined by histopathologic assessment of the resection specimen. The R0 resection rate will be analyzed among all eligible patients, including those not resected due to early progression, death or off-study.

SECONDARY OUTCOMES:
Progression-free survival | From randomization until the time of progression or death, up to approximately 6 years
  Progression-free survival is defined as the time from the date of randomization (or registration on Arm 4) to first objective documentation of progressive disease (distant or local) or death. Disease status is evaluated using RECIST (Response Evaluation Criteria in Solid Tumors). Disease progression is defined as having at least a 20% increase in the sum of the longest diameter (LD) of target lesion, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Overall survival | From randomization until the time of death, up to approximately 6 years
  Overall Survival (OS) is defined as the time from randomization (or registration on Arm 4) to death due to any cause, or censored at date last known alive.
Pathologic complete response | Up to 8 months after baseline
  The proportion of participants that achieved a pathologic complete response. Pathologic complete response is defined as the disappearance of all target lesions, as confirmed by a pathologist evaluating the tissue samples removed during surgery.
Number of participants with treatment related serious adverse events | From the start of treatment until 30 days after the end of treatment, up to approximately 14 months
  Adverse events are assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Adverse events are considered to be related to treatment if the Investigator deems them to be either possibly, probably, or definitely related to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Y. Wo, MD, Principal Investigator — Massachusetts General Hospital
Locations (10):
- United States (10):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Newton Wellesley Hospital, Newton, Massachusetts
  - New York University Langone Medical Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang H, Yuan S, Wang H. Current Status of Research on Losartan in Tumour Therapy. J Cell Mol Med. 2026 Jan;30(1):e70985. doi: 10.1111/jcmm.70985. PMID 41486497